CLINICAL TRIAL: NCT02296333
Title: Double Blinded Study Ondansetron's Opposite Effect on Postoperative Analgesia of Acetaminophen
Brief Title: Ondansetron's Opposite Effect on Postoperative Analgesia of Acetaminophen
Acronym: OOEOPAOA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Onur Koyuncu, Assistant Proffesor, Mustafa Kemal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 03 2014 05
Record Dates: First submitted 2014-08-24; First posted 2014-11-20 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2015-03

CONDITIONS: Postoperative Pain
Keywords: Acetaminophen, ondansetron
MeSH Terms: conditions — Pain, Postoperative | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ondansetron (Active Comparator): ondansetron iv, 8 mg, skin closure time
  Interventions: Drug: ondansetron
- isotonic (Placebo Comparator): isotonic 2ml, once, skin closure time
  Interventions: Drug: isotonic

INTERVENTIONS:
Drug: ondansetron — 8 mg intravenous in the skin closure
  Other Names: Zofran
  Arms: ondansetron
Drug: isotonic — 8 mg intravenous in the skin closure
  Arms: isotonic

SUMMARY:
The purpose of the study is to determine whether the effect of ondansetron on the analgesic effect of acetaminophen. Because 5HT3 blockers prevent the analgesic effects of acetaminophen and also reduce opioid consumption

DETAILED DESCRIPTION:
The investigators enrolled 80 American Society of Anesthesiologists Physical Status I-II women 18-80 years old scheduled for hysterectomy under general anesthesia over the course of a year. The study will be restricted hysterectomies with horizontal abdominal skin incision who will be able to operate a patient-controlled analgesia (PCA) device.

Participating women will be premedicated with 1-2 mg intravenous (IV) midazolam per preference of the attending anesthesiologist.

Anesthesia will be induced with propofol (2 mg/kg IV); intubation will be facilitated by rocuronium (0.6 mg/kg IV); and anesthesia will be maintained by sevoflurane in combination with nitrous oxide 50% in oxygen. Fentanyl, 2 µg/kg intravenous will be given 3-5 min before the surgical incision.

After endotracheal intubation, all patients' lungs will be mechanically ventilated to maintain the end-expiratory carbon dioxide values between 34 and 36 mmHg.

A Pfannenstiel approach will be used in each woman, and the same surgeon will be conducted all operations.

Randomization will be web-based and out of the control of any investigator. The web system will be accessed by the anesthesia resident at the induction. Drugs will be covered by opaque plastic to keep the surgical team and anesthesiologists blinded to treatment.

Both groups patients will be received 1 g acetaminophen in 100 ml saline given every 6 hours starting with the skin closure for 24 hours, an amount generally regarded as safe.

1. Group I patients will be received '8 mg ondansetron hydrochloride'
2. Group II patients will be received '2 ml saline' Both of them will be applied in a 100 ml saline bag at the same time with the skin closure.

After return of spontaneous ventilation and tracheal extubation, patients will be transferred to the post anesthesia care unit (PACU).

Patients were connected to a patient-controlled analgesia (PCA) device and postoperative analgesia will be provided using 20-mg intravenous bolus injections of tramadol at a lockout interval of 15 min and with a maximum 4-h limit of 150 mg. The PCA device will be discontinued when the patient made no demands for the opioid analgesic in the preceding 4-h interval or at a maximum of 24 hours after surgery.

* heart rate
* systolic arterial blood pressures
* diastolic arterial blood pressures
* mean arterial blood pressures
* oxygen saturation
* respiratory rate
* visual analogue scales while sitting and laying
* tramadol consumption
* additive analgesics
* complications
* postoperative nausea and vomiting scores
* antiemetic use will be assessed at PACU, 1th. hour, 4th hour, 8th hour, 12th hour, 16th hour, 20th hour and 24th hour.
* Pain satisfaction scale
* ambulation time
* first flatus time
* oral intake time
* Hospital anxiety and depression scale

When pain scores were VAS ≥5, then as a rescue analgesics 75 mg diclofenac Na intramuscularly will be given. If systolic arterial pressure (SAP) will be <90 mmHg or mean arterial pressure will be <50 mmHg, 5 mg intravenous ephedrine HCl will be given. If the heart rate will be <50 beats/minute, 0.5 mg atropine sulfate intravenous will be given. When patients sustained nausea or vomiting lasting longer than 5 minutes, metoclopramide (10 mg intravenously) will be given.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-80 years old scheduled for hysterectomy
* Horizontal or vertical abdominal skin incision
* Ability to operate a patient-controlled analgesia (PCA) device
* Written informed consent.

Exclusion Criteria:

* Emergency or urgent procedures
* Women with pre-existing chronic pain at any site requiring opioid analgesia
* Who had a history of significant Axis I psychiatric disease (major depressive disorder, bipolar disorder, schizophrenia, etc.)
* Significant hepatic (alanine aminotransferase or aspartate aminotransferase >2 times normal) or renal (serum creatinine >2 mg/dl) impairment
* Allergy to ondansetron or acetaminophen
* Were pregnant

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-05; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | Postoperative 24 hours
  Visual analogue scale
Opioid (tramadol) consumption | Postoperative 24 hours
  Tramadol consumption

SECONDARY OUTCOMES:
Postoperative complications | Postoperative 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Onur Koyuncu, Ass.prof, Study Chair — Mustafa Kemal University Medicine Faculty
Locations (1):
- Mustafa Kemal University Medicine Faculty, Hatay, Turkey (Türkiye)

REFERENCES:
- [Result] Tjolsen A, Lund A, Hole K. Antinociceptive effect of paracetamol in rats is partly dependent on spinal serotonergic systems. Eur J Pharmacol. 1991 Feb 7;193(2):193-201. doi: 10.1016/0014-2999(91)90036-p. PMID 1904822
- [Result] Pickering G, Loriot MA, Libert F, Eschalier A, Beaune P, Dubray C. Analgesic effect of acetaminophen in humans: first evidence of a central serotonergic mechanism. Clin Pharmacol Ther. 2006 Apr;79(4):371-8. doi: 10.1016/j.clpt.2005.12.307. PMID 16580905
- [Result] Jokela R, Ahonen J, Seitsonen E, Marjakangas P, Korttila K. The influence of ondansetron on the analgesic effect of acetaminophen after laparoscopic hysterectomy. Clin Pharmacol Ther. 2010 Jun;87(6):672-8. doi: 10.1038/clpt.2009.281. Epub 2010 Mar 10. PMID 20220746
- See also: http://www.ncbi.nlm.nih.gov/pubmed/20220746 — http://www.ncbi.nlm.nih.gov/pubmed/20220746